CLINICAL TRIAL: NCT00003574
Title: A Multi-Center, Open-Label Clinical Study to Evaluate the Safety and Performance of the Proxima GliaSite RTS, a Radiation Delivery System, in Patients With Recurrent Malignant Brain Tumors Undergoing Surgical Resection
Brief Title: Radiation Therapy in Treating Patients With Progressive or Recurrent Malignant Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066641; NABTT-9801; JHOC-NABTT-9801
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2000-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Surgical Procedures, Operative; Brachytherapy; Iodine-125

INTERVENTIONS:
Procedure: surgical procedure
Radiation: brachytherapy
Radiation: intraoperative radiation therapy
Radiation: iodine I 125

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy in treating patients who are undergoing surgical removal of progressive or recurrent malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety of the GliaSite RTS in patients with progressive or recurrent malignant brain tumors undergoing surgical resection. II. Evaluate the performance of the GliaSite RTS in these patients.

OUTLINE: This is an open label, multicenter study. Patients undergo surgical resection of the tumor followed by surgical placement of the GliaSite device in the resection cavity. One to 2 weeks after surgery, patients receive brachytherapy consisting of an infusion of iodine I-125. The I-125 solution is removed and collected 5-7 days later. The device is surgically removed within 24 hours. Patients are followed at 24 hours, 14 days, and 1 year post device removal.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant glioma: Anaplastic astrocytoma Anaplastic oligodendroglioma Glioblastoma multiforme Unifocal disease Progressive or recurrent disease following radiation therapy and/or chemotherapy Must be eligible for surgical resection of the tumor mass No unresectable leptomeningeal spread or ventricular invasion outside the radiation treatment volume No exophytic ventricular tumors Must have a maximal cross-sectional diameter enhancing tumor greater than 2.0 cm but not greater than 5.0 cm by preoperative MRI Ratio of major axes of the tumor should not exceed 1.5 No marked edema by preoperative MRI or CT that cannot be corrected by tumor resection

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No uncontrolled hypertension, angina pectoris, or uncontrolled cardiac dysrhythmia Other: Not pregnant or nursing Fertile patients must use effective contraception No serious concurrent infection or other medical illness No prior or concurrent malignancy within 5 years except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: See Disease Characteristics No concurrent chemotherapy At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas) and recovered Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 months since prior radiotherapy and recovered Surgery: See Disease Characteristics Other: At least 4 weeks since prior use of medical device No concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tatter, MD, PhD, Study Chair — Wake Forest University Health Sciences
Locations (9):
- United States (9):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas